CLINICAL TRIAL: NCT03848026
Title: The Relationship Between the Tympanostomy Tube Extrusion Time & Viscosity
Brief Title: Tympanostomy Tube Extrusion Time & Viscosity
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Nazan Degirmenci, Principal Investigator, Bezmialem Vakif University
Other Study IDs: B.30.2.BAV.0.05.05/468
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: OTITIS MEDIA WITH EFFUSION
Keywords: Otitis media; tympanostomy tube; viscosity; middle ear fluid
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: middle ear fluid viscosity <439 centipoise (cP), Tympanostomy tube extrusion time of the all patients recorded prospectively
  Interventions: Other: Middle ear fluid viscosity; Other: Tympanostomy tube extrusion time
- Group 2: middle ear fluid viscosity >439 centipoise (cP), Tympanostomy tube extrusion time of the all patients recorded prospectively
  Interventions: Other: Middle ear fluid viscosity; Other: Tympanostomy tube extrusion time

INTERVENTIONS:
Other: Middle ear fluid viscosity — The patients were subdivided into two groups according to median viscosity level
Other: Tympanostomy tube extrusion time — Tympanostomy tube extrusion time of the all patients recorded prospectively.

SUMMARY:
Studies have focused on the factors that influence tympanostomy tube (TT) extrusion may contribute to the management of OME. In this study the investigators aimed to assess the correlation between the TT extrusion time and viscosity of the middle ear fluid. 33 patients scheduled for TT insertion included in the study. During the paracentesis, fluid from the middle ear was obtained, and the viscosity was measured with a viscometer. After the surgery, patients were controlled monthly until the tubes were seen extruded.The analysis of the correlation between tube extrusion time and viscosity was insignificant (p >0.05).

DETAILED DESCRIPTION:
45 patients were evaluated in the outpatient clinic of the Bezmialem Vakif University Department of Otorhinolaryngology. OME was diagnosed by endoscopic-otoscopic examination findings and type-B tympanograms. Patients who do not have a previous history of TT insertion and retraction pocket included in the study. They were all scheduled for Shepard TT insertion. 12 patients were excluded for not coming to their postoperative controls properly. Total of 33 patients' data were analyzed in the end. During the paracentesis, myringotomy incision was done at the anteroinferior quadrant. Fluid from the middle ear was obtained by using 22 gauge syringe, and the viscosity was measured with a viscometer. Since the viscosity in most patients was mucoid in appearance, the patients were subdivided into two groups according to median viscosity level to determine whether higher or lower viscosity of the effusion impacted tympanostomy tube extrusion time. Patients with an effusion below and above the median viscosity value of 439 centipoise (cP) were assigned to Group 1 and 2, respectively. After the surgery, patients were controlled monthly until the tubes were seen extruded.Brookfield DV-II+ProCP Viscometer (Brookfield Engineering Laboratories, Inc., Massachusetts, USA) was used for viscosity measurements. This viscometer was able to measure the viscosity of fluid samples as small as 0.5 ml. The results of the viscosity measurements were recorded as cP units. The patients were investigated for any correlation between the viscosity level of the effusion and extrusion time of the TT. Descriptive statistics were presented as mean and standard deviation. T-test was used to estimate the correlation between the parameters. Mann-Whitney U Test was used to compare the two groups. Statistical analyses were conducted with the IBM SSPS 22.0 program. Significance level was set at 0.05 for all tests. All the procedures were approved and performed in accordance with the ethical standards of the relevant national and institutional guidelines on human experimentation and with the Helsinki Declaration of 1975, as revised in 2008. Permission for the study was obtained from Institutional Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* endoscopic-otoscopic examination findings of serous otitis media
* type-B tympanograms
* None existence of a previous history of TT insertion
* None existence of a retraction pocket

Exclusion Criteria:

* Patients who do not come to their postoperative controls
* existence of a previous history of TT insertion
* existence of a retraction pocket

Ages: 2 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 33 patients who were diagnosed as otitis media with effusion and scheduled for Shepard TT insertion included in the study.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Mean tube extrusion time | 2 year
  Mean tube extrusion time of total 33 patients was measured
The correlation between tube extrusion time and viscosity | 2 year
  The correlation between tube extrusion time and viscosity was analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Degirmenci, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Degirmenci N, Tugrul S, Goktas SS, Senturk E, Calim OF, Dogan R, Yenigun A, Ozturan O. The relationship between the tympanostomy tube extrusion time and viscosity. Int J Pediatr Otorhinolaryngol. 2020 Sep;136:110140. doi: 10.1016/j.ijporl.2020.110140. Epub 2020 May 27. PMID 32554135